CLINICAL TRIAL: NCT06426498
Title: Developing a Method of Adjusting the Strength of Transcranial Focused Ultrasound (tFUS) to Personalize Treatment.
Brief Title: tFUS Induced Transient Scotoma for Individual Dosing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Mark George, Professor-Faculty, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00132894
Record Dates: First submitted 2024-05-14; First posted 2024-05-23 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Healthy
Keywords: ulltrasound; tFUS; scotoma; visual field
MeSH Terms: conditions — Scotoma

STUDY DESIGN:
Masking Description: The device will be on either right or left V1, and the ultrasound will be cycling on or off during the session. Subjects and investigators will be masked to on/off timing and puck location.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- tFUS over V1 (Experimental): All subjects will get tFUS, open label
  Interventions: Device: Brainsonix Bx Pulsar machine tFUS

INTERVENTIONS:
Device: Brainsonix Bx Pulsar machine tFUS — This is a tFUS device, delivering ultrasound at a dose within the FDA safety guidelines.

SUMMARY:
The purposes of this research study is to:

1. Develop a technique of transcranial Focused Ultrasound Stimulation (tFUS) where meaningful effects on the brain can be easily measured.
2. Use this technique to measure threshold for effective tFUS in individuals.
3. Determine whether disruption of conscious visual detection, versus non-conscious visually-guided behavior have different thresholds for disruption with tFUS.

DETAILED DESCRIPTION:
Transcranial focused ultrasound (tFUS) is a new noninvasive way to stimulate the brain in an awake and alert person. Investigators do not yet have an easily observable way to know whether they are in the right brain location with the correct dose for that person. Investigators wonder if they can produce a transient change in someone's visual field, called a scotoma, and whether they can use that to determine the minimum tFUS dose for that person.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18-70
* Normal or corrected-to normal vision and hearing
* No neurological or psychological illness

Exclusion Criteria:

* Diagnosis of any depressive or anxiety disorder
* Diagnosis of schizophrenia or bipolar disorder
* Current use of any non-prescribed psychoactive medications or drugs
* Contraindication to enter the MRI environment.
* Pregnancy (or suspected/possible pregnancy or plan to become pregnant in the short term).
* Urine Pregnancy Test: If the subject is a woman of childbearing potential and /or a man capable of fathering a child before, during, and/or after participation precaution should be taken. Examples of acceptable methods of birth control for participants involved in the study include: birth control pills, patch, IUD, condom, sponge, diaphragm with spermicide, or avoiding sexual activity that could cause the subject to become pregnant.
* Inability to adhere to treatment schedule.
* Initiation of new antidepressant treatment at the time of study randomization.

NOTE: There will be no exclusion based upon gender or minority status. We anticipate that at least 50% of the participants will be women. The percentage of minority participants is expected to be at least 5%. We will make vigorous attempts to increase this number by posting advertisement flyers in minority communities.

Children, prisoners, and institutionalized individuals will not be recruited, because they are beyond the scope of the objectives. Moreover, we will emphasize that participation in this study is completely voluntary. Recruitment of women and minorities has been addressed above. Non-English speaking subjects will not be recruited because they may not be able to understand instructions, which could undermine the validity of the results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2026-05-20 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Temporary Scotoma | During and immediately after (10 minutes) the tFUS
  Production of a temporary Scotoma as assessed by visual field testing of briefly presented objects in different quadrants while staring at a central cross on a computer screen.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina Brain Stimulation Division, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No